CLINICAL TRIAL: NCT06483633
Title: Effects of Combining Different Exercise Modes With Cold Pressor Test on Vascular Function and Sleep Quality in Female University Students With Sleep Disorders
Brief Title: Effects of Combining Different Exercise Modes With CPT on Vascular Function and Sleep Quality in Female University Students With SD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Sport University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: EOCDEMWCPTOVFASQIFUSWSD
Record Dates: First submitted 2024-06-23; First posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Sleep Quality; Vascular Function
Keywords: exercise; sleep disorders; cold pressor test; vascular function
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Motor Activity; Sleep Wake Disorders | interventions — 2-cyclohexylidenhydrazo-4-phenyl-thiazole

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- sleep disorder group (Experimental)
  Interventions: Behavioral: MICT + CPT, HIIT + CPT, SIT + CPT
- Control group (Experimental)
  Interventions: Behavioral: MICT + CPT, HIIT + CPT, SIT + CPT

INTERVENTIONS:
Behavioral: MICT + CPT, HIIT + CPT, SIT + CPT — Single acute intervention, each exercise mode had a washout period of at least 7 days.

SUMMARY:
Fourteen female college students with sleep disorders (SD) and fourteen with good sleep status were recruited, divided into sleep disorder group (SDG) and control group (CG). Both groups underwent moderate-intensity continuous training (MICT), high-intensity interval training (HIIT), and sprint interval training (SIT). Immediately after exercise, Cold Pressor Test (CPT) was administered, vascular indicators were measured immediately and 30 minutes later. The next day after exercise, participants completed the Pittsburgh sleep quality index (PSQI). Each exercise mode had a washout period of at least 7 days.

DETAILED DESCRIPTION:
Both SDG and CG underwent HIIT, MICT, and SIT interventions. After the exercise, a CPT was conducted, and vascular indicators were immediately measured at the end of the intervention. Another measurement was taken 30 minutes after the intervention. The exercise was performed on a power bike, with the requirement to maintain a pedaling frequency of 60 rpm. The exercise protocols for HIIT, MICT, and SIT were designed with equal exercise volume. The HIIT protocol consisted of 4 sets of 4 minutes at 85% maximal oxygen uptake data (VO2max), interspersed with 3 minutes at 50% VO2max. The MICT protocol involved continuous pedaling at 60% VO2max for 32 minutes. The SIT protocol included 6 sets of 30-second all-out sprints (100% VO2max) with 4.5 minutes of recovery at 60% VO2max between each sprint. There was a minimum of 7 days between each exercise mode as a washout period. The PSQI questionnaire was completed the day after each intervention upon waking up.

ELIGIBILITY:
Inclusion Criteria:

* Female university students aged between 18 and 30 years old
* Body Mass Index (BMI) between 18.5~24.0 kg/m2
* Presence of SD (PSQI > 8 points) or good sleep quality (PSQI ≤ 7 points)
* Not taking medications that affect sleep
* No cardiovascular diseases
* No regular exercise habits or specialized training but possessing the ability to complete the exercise program

Exclusion Criteria:

* Severe organic diseases such as heart, kidney, etc
* Metabolic diseases such as diabetes, etc.
* Taking medications that affect sleep (including drugs that promote or interfere with sleep)
* Permanent and severe exercise dysfunction
* Participation in other experiments

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Pittsburgh Sleep Quality Index | The next morning following each intervention, within 24 hours post-intervention
  The change of Pittsburgh Sleep Quality Index (PSQI) before and after the intervention, Pittsburgh Sleep Quality Index include: specifically PSQI total score, sleep quality, sleep latency, sleep duration, sleep efficiency, sleep disturbances, and daytime functioning.
Ankle-brachial pulse wave velocity (baPWV) | Immediately after each intervention and 30 minutes later.
  The change of baPWV before and after intervention.
Ankle-brachial index (ABI) | Immediately after each intervention and 30 minutes later.
  The change of ABI before and after intervention.

SECONDARY OUTCOMES:
Blood pressure | Immediately after each intervention and 30 minutes later.
  The change of blood pressure before and after intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- School of Sports Medicine and Rehabilitation, Beijing Sport University, Beijing, China